CLINICAL TRIAL: NCT05027594
Title: A Phase I Dose Escalation Study of NMS-03597812, a PERK Inhibitor, in Adult Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Ph I Study in Adult Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision is not based on emerging safety or efficacy concerns but on strategic reasons related to the changing and competitive treatment options in Multiple Myeloma
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PERKA-812-001; 2020-004351-32 (EudraCT Number)
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
Keywords: Phase I; Multiple Myeloma; PERK inhibitor
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase 1 Dose escalation part followed by a Dose Expansion part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Part (Experimental): Patients with a confirmed diagnosis of relapsed or relapsed and refractory multiple myeloma (as per IMWG criteria) who have exhausted standard treatment options that are expected to provide meaningful clinical benefit or for whom standard therapy is considered unsuitable
  Interventions: Drug: NMS-03597812
- Dose Expansion Part - NMS-03597812 single agent (Experimental): Patients with a confirmed diagnosis of relapsed or relapsed and refractory multiple myeloma (as per IMWG criteria) who have exhausted standard treatment options that are expected to provide meaningful clinical benefit or for whom standard therapy is considered unsuitable
  Interventions: Drug: NMS-03597812
- Dose Expansion Part - NMS-03597812 in combination with dexamethasone (Experimental): Patients with a confirmed diagnosis of relapsed or relapsed and refractory multiple myeloma (as per IMWG criteria) who have exhausted standard treatment options that are expected to provide meaningful clinical benefit or for whom standard therapy is considered unsuitable
  Interventions: Drug: NMS-03597812 + dexamethasone

INTERVENTIONS:
Drug: NMS-03597812 — All patients will receive NMS-03597812 administered orally once daily on Days 1-21 in repeated 4-week cycles.
  Arms: Dose Escalation Part; Dose Expansion Part - NMS-03597812 single agent
Drug: NMS-03597812 + dexamethasone — All patients will receive NMS-03597812 administered orally once daily on Days 1-21 and Dexamethasone administered orally once a week on Days 1, 8, 15 and 22 in repeated 4-week cycles.
  Arms: Dose Expansion Part - NMS-03597812 in combination with dexamethasone

SUMMARY:
This is a Phase I, first-in-human (FIH), open-label, non-randomized, multi-center study to explore the safety, tolerability, pharmacokinetics and preliminary antitumor activity of NMS-03597812 in adult patients with RRMM who have exhausted standard treatment options that are expected to provide meaningful clinical benefit or for whom standard therapy is considered unsuitable.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis of relapsed or relapsed and refractory multiple myeloma (as per IMWG criteria)
2. Patients must have exhausted available therapeutic options that are expected to provide meaningful clinical benefit, either through disease relapse, treatment refractory disease, intolerance or refusal of the therapy.
3. Patients must have received at least three prior lines of therapy as defined by IMWG, including a proteasome inhibitor, an immunomodulatory agent, and an anti-CD38 antibody.
4. Patients must have progressive/refractory disease to the last line of therapy.
5. Patients must have measurable disease, defined as any of the following:serum monoclonal protein ≥ 0.5 g/dL by protein electrophoresis, ≥200 mg of monoclonal protein in urine on 24-h electrophoresis, or serum immunoglobulin free light chain ≥10 mg/dL with abnormal free-light-chain ratio.
6. Adult (age ≥18 years) patients.
7. Karnofsky performance status ≥60%.
8. All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to NCI CTCAE version 5.0 Grade ≤1 or according to inclusion criterion 9.
9. Adequate hematological profile, renal, hepatic and pancreatic functions
10. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within the screening period prior to start of the study drug.
11. Patients must use effective contraception or abstinence. Female patients of childbearing potential must agree to use effective contraception or abstinence during the period of therapy and in the following 90 days after discontinuation of study treatment. Male patients must be surgically sterile or must agree to use effective contraception or abstinence during the period of therapy and in the following 90 days after discontinuation of study treatment.
12. Ability to swallow capsules intact (without chewing, crushing, or opening).
13. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study indications or procedures.
14. Signed and dated IRB/EC-approved Informed Consent

Exclusion Criteria:

1. Current enrollment in another interventional clinical study.
2. Diagnosis of primary refractory multiple myeloma defined as disease that is non-responsive in patients who have never achieved a minimal response or better with any therapy
3. Diagnosis of plasma cell leukemia, Waldenstrom's macroglobulinemia or amyloidosis.
4. Diagnosis of non-secretory myeloma.
5. Known central nervous system (CNS) involvement by multiple myeloma.
6. Known history of polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes (POEMS) syndrome.
7. Currently active second malignancy, except for adequately treated basal or squamous cell skin cancer and/or conebiopsied in situ carcinoma of the cervix uteri and/or superficial bladder cancer.
8. Autologous stem cell transplant ≤3 months prior to starting NMS-03597812.
9. Prior allogeneic hematopoietic stem cell transplant (HSCT) with either standard or reduced intensity conditioning ≤6 months prior to starting NMS-03597812.
10. Active acute or chronic graft versus host disease (GVHD) requiring immunosuppressive treatment. Patients who experienced GVHD requiring immunosuppressive treatment, must have stopped immunosuppressive treatment >3 months prior to starting NMS-03597812.
11. Any anticancer agent within 3 weeks (6 weeks for immunotherapy or nitrosoureas).
12. Prior CAR-T cell <3 months prior to starting NMS-03597812.
13. Concomitant oral prednisone(or equivalent)>10 mg/day. Doses of corticosteroid must have been stable for at least 7 days before startingNMS-03597812.
14. Major surgery within 4 weeks before treatment start.
15. Radiotherapy within 3 weeks prior to starting NMS-03597812. However, if the radiation portal covered ≤ 5% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy.
16. Patient with evidence of clinically significant mucosal or internal bleeding.
17. Patient platelet transfusion refractory.
18. History of pancreatitis or current alcohol abuse.
19. Uncontrolled diabetes.
20. Patients with QTc interval ≥ 480 milliseconds or with risk factors for torsade de pointes (e.g., uncontrolled heart failure, uncontrolled hypokalemia, history of prolonged QTc interval or family history of long QT syndrome). For patients receiving treatment with concomitant medications known to prolong the QTc interval, replacement with another treatment should be considered. If replacement or discontinuation is not clinically feasible, a careful risk/benefit evaluation should be performed prior to enrollment.
21. Breast-feeding or planning to breast feed during the study or within 3 months after study treatment.
22. Known hypersensitivity to any of the components of the NMS-03597812 drug product.
23. Known hypersensitivity to steroids or any of the components of the dexamethasone drug product (applies only to the expansion cohort testing NMS-03597812 in combination with dexamethasone).
24. Any of the following in the previous 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
25. Uncontrolled bacterial, viral, or fungal infections including: known infection with HIV, HBV and/or HCV; patients who are seropositive following HBV vaccine are eligible.
26. Known active gastrointestinal disease (e.g., documented gastrointestinal ulcer, Crohn's disease, ulcerative colitis or short gut syndrome) or other malabsorption syndromes that would impact drug absorption or represent a contra-indication for the treatment with dexamethasone (NMS-03597812 and dexamethasone expansion cohort).
27. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study or could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
28. Patient who are receiving concomitant medications that are strong inducers or inhibitors of CYP34A and CYP2C9 that cannot be replaced with alternative therapy.
29. Patients who are receiving concomitant medications that are sensitive substrates of CYP3A4 and CYP2D6 with narrow therapeutic window that cannot be replaced with alternative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with first-cycle dose limiting toxicity | Time interval between the date of the first dose administration in Cycle 1 (each cycle is 28 days) and the date of the first dose administration in Cycle 2 which is expected to be 28 days or up to 42 days in case of dose delay due to toxicity
  For DLT evaluation, severity (grade) is classified according to common terminology criteria for adverse events version 5.0 (CTCAE v5.0).

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From the Informed Consent signature to 28 days after the last dose of study treatment administration
  Safety will be assessed by adverse events (AEs), which include clinically significant abnormalities identified during a medical test (e.g. laboratory tests, electrocardiogram, vital signs, physical examinations). AEs will be coded by Medical Dictionary for Regulatory Activities (MedDRA) and their severity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). The analysis will focus on the events reported after the start of treatment (treatment emergent adverse events).
Number of Participants by Best Tumor response | From treatment start date until disease progression or relapse (up to approximately 12 months).
  Number of patients with best tumor response achieved on treatment is determined using International Myeloma Working Group (IMWG) Criteria 2016. The number of patients is provided for each category: Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), Minimal Response (MR), Stable Disease (SD), Progressive Disease (PD) and Not Evaluable (NE).
Number of Participants with Overall Response | From treatment start date until disease progression or relapse (up to approximately 12 months).
  Best Overall Response is measured for patients achieving Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR) or Partial Response (PR) as Best Response according to International Myeloma Working Group (IMWG) Criteria 2016
Number of Participants with Clinical Benefit | From treatment start date until disease progression or relapse (up to approximately 12 months).
  Clinical Benefit is measured for patients achieving Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR) or Minimal Response (MR) as Best Response according to International Myeloma Working Group (IMWG) Criteria 2016.
Duration of Response | From the first responding tumor assessment until Progression Disease/Relapse or Death due to Progression (up to approximately 12 months)
  Duration of Response is calculated in patients achieving overall response by International Myeloma Working Group (IMWG) Criteria 2016, as the time elapsed from the date at which Overall response is first observed to the date of first observed disease progression/relapse or date of death due to progression, whichever comes first
Progression Free Survival (PFS) | From date of first dose of study drug up to the date of first documentation of disease progression/relapse or death due to any cause, whichever comes first (up to approximately 12 months).
  Progression Free Survival (PFS) is calculated as the time elapsed from the date of treatment initiation to the date of first documentation of disease progression/relapse according to International Myeloma Working Group (IMWG) Criteria 2016, or death due to any cause, whichever comes first
Maximum concentration (Cmax) of NMS-03597812 after single and multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and at Cycle 2 on Days 1, 8, 15, 21 at different timepoints.
  Plasma samples will be collected and used for pharmacokinetics assessments.
Time to maximum plasma concentration (Tmax) of NMS-03597812 after single and multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and at Cycle 2 on Days 1, 8, 15, 21, at different timepoints.
  Plasma samples will be collected and used for pharmacokinetics assessments.
Area under the plasma concentration versus time curve up to the last detectable plasma concentration (AUClast) of NMS-03597812 after single and multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and at Cycle 2 on Days 1, 8, 15, 21, at different timepoints.
  Plasma samples will be collected and used for pharmacokinetics assessments.
Minimum plasma concentration (Cmin) of NMS-03597812 after single and multiple doses of drug. | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and at Cycle 2 on Days 1, 8, 15, 21, at different timepoints.
  Plasma samples will be collected and used for pharmacokinetics assessments.
Average plasma concentration (Cave) of NMS-03597812 after multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and at Cycle 2 on Days 1, 8, 15, 21, at different timepoints.
  Plasma samples will be collected and used for pharmacokinetics assessments
Area under the plasma concentration versus time curve to infinity (AUCinf) of NMS-03597812 after multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and Cycle 2 on Days 1, 8, 15, 21 at different timepoints.
  Plasma samples will be collected and used for pharmacokinetics assessments.
Terminal elimination half-life (t1/2) of NMS-03597812 after multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and Cycle 2 on Days 1, 8, 15, 21, at different timepoints
  Plasma samples will be collected and used for pharmacokinetics assessments
Oral plasma clearance (CL/F) of NMS-03597812 after multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and at Cycle 2 on Days 1, 8, 15, 21, at different timepoints.
  Plasma samples will be collected and used for pharmacokinetics assessments.
Apparent volume of distribution (Vd/F) of NMS-03597812 after multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and at Cycle 2 on Days 1, 8, 15, 21, at different timepoints
  Plasma samples will be collected and used for pharmacokinetics assessments.
Accumulation ratio (Rac) of NMS-03597812 after multiple doses of drug | At Cycle 1 (each cycle is 28 days) on Days 1, 2, 8, 15, 21, 22, 23 and 24 and at Cycle 2 on Days 1, 8, 15, 21, at different timepoints
  Plasma samples will be collected and used for pharmacokinetics assessments.
Renal clearance of NMS-03597812 after multiple doses of drug. | At Cycle 1 (each cycle is 28 days) Day 1 and Day 21
  Urine samples will be used for PK assessments. Samples will be collected in patients treated in the dose escalation phase, starting from cohort 4 or from the occurrence of the first DLT, whichever comes first, and in all patients treated in the dose expansion.
Cumulative amount recovered unchanged in the urine (Ae) of NMS-03597812 after multiple doses of drug | At Cycle 1 (each cycle is 28 days) Day 1 and Day 21
  Urine samples will be used for PK assessments. Samples will be collected in patients treated in the dose escalation phase, starting from cohort 4 or from the occurrence of the first DLT, whichever comes first, and in all patients treated in the dose expansion.
Cumulative amount recovered unchanged in the urine expressed as a fraction of administered dose (Ae%) of NMS-03597812 after multiple doses of drug. | At Cycle 1 (each cycle is 28 days) Day 1 and Day 21
  Urine samples will be used for PK assessments. Samples will be collected in patients treated in the dose escalation phase, starting from cohort 4 or from the occurrence of the first DLT, whichever comes first, and in all patients treated in the dose expansion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dana- Farber Cancer Institute, Boston, Massachusetts
  - Levine Cancer Institute, Charlotte, North Carolina